CLINICAL TRIAL: NCT04308486
Title: Anti-mullerian Hormone,Testesterone,Esrtadiol,Testesterone/Esrtadiol Ratio as Predictive Values for TESA and TESE Outcome in Non Obstructive Azoospermia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Ahmed Ashraf Fakhr Eldeen Hamoda, Doctor, Assiut University
Other Study IDs: prediction of TESA and TESE
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Non-obstructive Azoospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
*Evaluate the predictive value of AMH, Testosterone,Estradiol,Testosterone Estradiol ratio for TESA and TESE outcome in non obstructive azoospermic patients.

DETAILED DESCRIPTION:
* The relevance of male infertility has progressively grown , with significant medical, psychological, and socio-economic implications. .. With no sperm found at multiple semen analyses, non-obstructive azoospermia (NOA) is the most severe form of infertility.
* The introduction to clinical practice of assisted reproduction techniques such as intra-cytoplasmic sperm injection (ICSI) made fatherhood possible for men with (NOA). The extraction of sperm from the testis through testicular sperm aspiration (TESA), testicular sperm extraction (TESE) or open biopsy can result in a favorable reproductive outcome. Nevertheless, all these procedures are invasive in nature with variable possibility of successful sperm extraction. As a consequence, a non-invasive test that could predict the presence of sperm in men with NOA would be of profound clinical importance
* However, the lack of useful predictive biomarkers suggestive for successful sperm retrieval at microTESE and TESA in NOA men still represents a relevant gap with a very negative return for the patient. Indeed, no significant association has been found between microTESEand TESA sperm retrieval outcomes and preoperative testicular volume, baseline follicular stimulating hormone (FSH) levels, basal level of Testosterone (T) or increased T level following treatments with aromatase inhibitors, clomiphene citrate or human chorionic gonadotropin.
* Therefore, it has been amust to identify novel and user-friendly prognostic factors reliably predicting surgical outcomes in NOA men in the real-life setting. Among other variables, some hormons can be subjected to studies for this purpose such as levels of testis-derived hormones (which might be representative of the primary testicular failure) as the Anti-Müllerian Hormone (AMH),( which is suggestive for a Sertoli cells' immature phenotype),and testosterone of biological relevance...
* An investigation from the early 1970s demonstrated that the human testis does indeed secrete estradiol within the spermatic vein, at amean concentration that is 50 times greater than that inthe peripheral plasma . These findings led to the hypothesis that local estrogen levels might be associated with the current stateof spermatogenesis, or the total number of spermatogenic cells in the testis.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of NOA associated with primary couple's infertility;
* age from 20 to 50 years old
* freedom from any known systemic diseases affecting the previous hormonal levels such as liver cirrhosis .
* hormonal therapy for at least two weeks prior to the surgery

Exclusion Criteria:

* obstructive azoospermia
* congenital bilateral absent vas

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 men within 20 to 50 years with non obstructive azoospermia undergoing TESA or TESE
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the predictive value of Anti-mullerian hormone,Testosterone,Estradiol,Testosterone/Estradiol ratio for TESA and TESE outcome in non obstructive azoospermia | baseline

REFERENCES:
- [Background] Alfano M, Ventimiglia E, Locatelli I, Capogrosso P, Cazzaniga W, Pederzoli F, Frego N, Matloob R, Sacca A, Pagliardini L, Vigano P, Zerbi P, Nebuloni M, Pontillo M, Montorsi F, Salonia A. Anti-Mullerian Hormone-to-Testosterone Ratio is Predictive of Positive Sperm Retrieval in Men with Idiopathic Non-Obstructive Azoospermia. Sci Rep. 2017 Dec 15;7(1):17638. doi: 10.1038/s41598-017-17420-z. PMID 29247212
- [Background] Matuszczak E, Hermanowicz A, Komarowska M, Debek W. Serum AMH in Physiology and Pathology of Male Gonads. Int J Endocrinol. 2013;2013:128907. doi: 10.1155/2013/128907. Epub 2013 Oct 24. PMID 24282408
- [Background] Toulis KA, Iliadou PK, Venetis CA, Tsametis C, Tarlatzis BC, Papadimas I, Goulis DG. Inhibin B and anti-Mullerian hormone as markers of persistent spermatogenesis in men with non-obstructive azoospermia: a meta-analysis of diagnostic accuracy studies. Hum Reprod Update. 2010 Nov-Dec;16(6):713-24. doi: 10.1093/humupd/dmq024. Epub 2010 Jul 1. PMID 20601364